CLINICAL TRIAL: NCT00689390
Title: Long-Term Follow-Up of Subjects in a Phase 1, 2, or 3 Clinical Trial in Which Boceprevir or Narlaprevir Was Administered for the Treatment of Chronic Hepatitis C
Brief Title: Three-year Follow-up of Participants After Administration of Boceprevir or Narlaprevir for the Treatment of Chronic Hepatitis C (P05063)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to satisfaction of post-marketing commitments
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P05063; 2006-006529-25 (EudraCT Number)
Record Dates: First submitted 2008-05-27; First posted 2008-06-03 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C, Chronic; Hepacivirus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; narlaprevir; peginterferon alfa-2b; Ribavirin; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Participants from Boceprevir Studies (Other): Participants who previously participated in treatment studies in which boceprevir was administered were subsequently enrolled in Part 1 of the current follow-up study P05063 (NCT00689390). Participants may have received boceprevir or control peginterferon plus ribavirin (PR) in the previous treatment study. No treatment was administered in the current follow-up study.
  Interventions: Biological: Boceprevir; Biological: Peginterferon alfa-2b; Drug: Ribavirin; Other: Blood/Plasma Collection
- Participants from Narlaprevir Studies (Other): Participants who previously participated in treatment studies in which narlaprevir was administered were subsequently enrolled in Part 2 of the current follow-up study P05063 (NCT00689390). Participants may have received narlaprevir or control PR in the previous treatment study. No treatment was administered in the current follow-up study.
  Interventions: Biological: Narlaprevir; Biological: Peginterferon alfa-2b; Drug: Ribavirin; Other: Blood/Plasma Collection

INTERVENTIONS:
Biological: Boceprevir — In previous treatment studies, boceprevir was administered as specified by the protocol. No treatment was administered on the current follow-up study (P05063, NCT00689390).
  Other Names: SCH 503034
  Arms: Participants from Boceprevir Studies
Biological: Narlaprevir — In previous treatment studies, narlaprevir was administered as specified by the protocol. No treatment was administered on the current follow-up study (P05063, NCT00689390).
  Other Names: SCH 900518
  Arms: Participants from Narlaprevir Studies
Biological: Peginterferon alfa-2b — In previous treatment studies, peginterferon alfa-2b was administered as specified by the protocol. No treatment was administered on the current follow-up study (P05063, NCT00689390).
  Other Names: PEG-Intron®; SCH 054031
Drug: Ribavirin — In previous treatment studies, ribavirin was administered as specified by the protocol. No treatment was administered on the current follow-up study (P05063, NCT00689390).
  Other Names: Rebetol®
Other: Blood/Plasma Collection — Blood samples were collected at all visits during the LTFU for blood chemistry and hematology. Plasma samples were collected at all visits as appropriate from participants who were sustained responders at the end of FU in the previous treatment protocol for HCV-RNA PCR and HCV sequence analysis.

SUMMARY:
Study P05063 is a 3-year long-term follow-up (LTFU) study in participants previously treated with boceprevir (BOC) or narlaprevir (NAR) in a Phase 1, 2, or 3 clinical study. Participants will be followed for up to 3.5 years after the end of their participation in the treatment protocol to document maintenance of the antiviral response (for sustained responders) and to characterize the long-term safety after use of this therapeutic regimen. LTFU procedures include collection of plasma samples for measuring Hepatitis C Virus ribonucleic acid (HCV-RNA) by polymerase chain reaction (PCR) and HCV sequence analysis. No drug therapy will be administered as part of this study.

DETAILED DESCRIPTION:
In Part 1, participants who previously participated in one of nine boceprevir studies (P03523 [NCT00423670], P03659 [NCT00160251], P04487 [No NCT], P05101 [NCT00708500], P05216 [NCT00705432], P05411 [NCT00959699], P05514 [NCT00910624], P05685 [NCT00845065], and P06086 [NCT01023035]) were followed for response. In Part 2, participants who previously participated in one narlaprevir study (P05104 [NCT00797745]) were followed for response.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing to give written informed consent and be able to adhere to the visit schedule.
* Participant must have received at least one dose of boceprevir or narlaprevir in a previous Phase 1, 2, or 3 clinical study.

Exclusion Criteria:

* Concurrent participation in any other clinical study for the treatment of chronic hepatitis C.
* Retreatment with any antiviral or immunomodulatory drug for chronic hepatitis C after completion of, or discontinuation from, the SPRI Phase 1, 2, or 3 clinical study in which the participant previously participated.
* Any condition which in the opinion of the Investigator would make the participant unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1954 (Actual)
Dates: Start 2007-02-20 (Actual); Primary Completion 2014-10-13 (Actual); Study Completion 2014-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Howe AY, Long J, Nickle D, Barnard R, Thompson S, Howe J, Alves K, Wahl J. Long-term follow-up of patients receiving boceprevir for treatment of chronic hepatitis C. Antiviral Res. 2015 Jan;113:71-8. doi: 10.1016/j.antiviral.2014.10.010. Epub 2014 Oct 24. PMID 25446895
- [Derived] Barnard R, Chopra A, James I, Blinco J, Watson MW, Jabara CB, Hazuda D, Lemon SM, Mallal S, Gaudieri S. Primer ID ultra-deep sequencing reveals dynamics of drug resistance-associated variants in breakthrough hepatitis C viruses: relevance to treatment outcome and resistance screening. Antivir Ther. 2016;21(7):567-577. doi: 10.3851/IMP3056. Epub 2016 May 24. PMID 27219495
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05063&kw=P05063&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 9 boceprevir studies (P03523 [NCT00423670], P03659 [NCT00160251], P04487 [No NCT], P05101 [NCT00708500], P05216 [NCT00705432], P05411 [NCT00959699], P05514 [NCT00910624], P05685 [NCT00845065], and P06086 [NCT01023035]) and 1 narlaprevir study (P05104 [NCT00797745]).
Pre-assignment Details: 1954 participants enrolled in this long-term follow-up (LTFU) study, with 1907 participants from 9 boceprevir studies and 47 participants from 1 narlaprevir study.
Period: Overall Study
Arm/Group | Participants From Boceprevir Studies | Participants From Narlaprevir Studies
Started | 1907 | 47
Completed | 1481 | 37
Not Completed | 426 | 10
Not completed — Adverse Event | 19 | 0
Not completed — Lost to Follow-up | 179 | 7
Not completed — Withdrawal by Subject | 117 | 3
Not completed — Withdrew Consent-Retreatment Opportunity | 52 | 0
Not completed — Non-Compliance With Protocol | 21 | 0
Not completed — Did Not Meet Protocol Eligibility | 1 | 0
Not completed — Administrative | 37 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants From Boceprevir Studies | Participants From Narlaprevir Studies | Total
Number analyzed (Participants) | 1907 | 47 | 1954
Age, Customized [Number; unit: participants]
  <40 years | 173 | 5 | 178
  40 to <65 years | 1651 | 42 | 1693
  ≥65 years | 83 | 0 | 83
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 785 | 19 | 804
  Male | 1122 | 28 | 1150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse During the LTFU Among Sustained Responders From Previous Treatment Studies With Boceprevir or Narlaprevir (Durability of Virologic Response)
Description: Durability of response was assessed by the number of participants who relapsed during the LTFU among those that had achieved sustained virologic response (SVR) by 24 weeks after treatment with boceprevir or narlaprevir in a previous Phase 1, 2, or 3 treatment study. In the current LTFU, participants were classified based on the last Hepatitis C Virus ribonucleic acid (HCV-RNA) result available at the time of the data cut-off date as follows: A participant was classified as a sustained virologic responder at a given time point if serum HCV-RNA was undetectable at that time point and there had not been a positive HCV-RNA since the participant was determined to have achieved SVR in the previous study. A participant was classified as a relapser if they were a sustained virologic responder in the previous treatment study and became serum HCV-RNA positive with no subsequent negative results during LTFU.
Time Frame: From End Of Treatment (EOT) date in the previous treatment study to the first date of a positive HCV RNA result for relapsers or the last contact date for non-relapsers in the LTFU (up to 3.5 years)
Population: All participants who were sustained responders at 24 weeks post-treatment in the previous study and who had available data were included in the analysis.
Measure: Number; unit: participants
Groups:
- Previous SVR on Boceprevir + PR: Participants who previously received boceprevir plus PR in treatment studies and achieved sustained virologic response (SVR). No treatment was administered in the current follow-up study.
- Previous SVR on Narlaprevir + PR: Participants who previously received narlaprevir plus PR in treatment studies and achieved SVR. No treatment was administered in the current follow-up study.
- Previous SVR on PR Only: Participants who previously received PR only in boceprevir or narlaprevir treatment studies and achieved SVR. No treatment was administered in the current follow-up study
Arm/Group | Previous SVR on Boceprevir + PR | Previous SVR on Narlaprevir + PR | Previous SVR on PR Only
Number analyzed (Participants) | 1116 | 40 | 144
participants | 8 | 0 | 1

2. Primary Outcome: Kaplan-Meier Exposure-adjusted Relapse Rate
Description: The distribution of time to relapse was summarized using Kaplan-Meier estimates for all participants who were sustained responders at 24 weeks post-treatment in the previous study. Exposure Adjusted Relapse Rate = 1000 × (number of relapses) / (Total exposure time in years). Total exposure time in years = [(total number of days from last day of treatment to the last follow-up day for all subjects who did not relapse) + (total number of days from last day of treatment to the day of relapse for those who relapsed)] / 365.25 days [for 1 year].
Time Frame: From EOT date in the previous treatment study to the first date of a positive HCV RNA result for relapsers or the last contact date for non-relapsers in the LTFU (up to 3.5 years)
Population: as for outcome 1
Measure: Number; unit: relapses per 1,000 person-years
Arm/Group | Previous SVR on Boceprevir + PR | Previous SVR on Narlaprevir + PR | Previous SVR on PR Only
Number analyzed (Participants) | 1116 | 40 | 144
relapses per 1,000 person-years | 2.3 | 0 | 2.2

3. Primary Outcome: Number of Participants With HCV Treatment-Emergent Resistance Associated Variants (TE-RAVs) of NS3/4A Protease Loci
Description: Plasma samples of all participants receiving at least one dose of study medication in a previous treatment protocol were evaluated by population sequencing and analyzed to detect amino acid variants in the NS3/4A protease known to be associated with reduced susceptibility to boceprevir and narlaprevir. RAVs in the NS3/4A protease gene were evaluated at 12 loci (V36, Q41, F43, T54, V55, V107, R155, A156, V158, D168, I/V170 and M175) on the basis of in vitro studies. A TE-RAV was defined as a RAV not present at baseline and that had not returned to wild type (WT) while the participant was still on treatment. The number of participants with TE-RAVS detected at the EOT in the previous treatment study are reported below, followed by those participants with TE-RAVS that returned to WT during the LTFU (among those with detected TE-RAVS).
Time Frame: From EOT in the previous treatment study to the last available date in the LTFU (up to 3.5 years)
Population: All participants with TE-RAVs who received at least one dose of study medication in a previous Phase 1, 2, or 3 boceprevir or narlaprevir clinical study. Participants could have had more than one TE-RAV. All TE-RAVs were observed in participants in the boceprevir studies (i.e. none of the participants in the narlaprevir study had a TE-RAV).
Measure: Number; unit: participants
Groups:
- Participants From Boceprevir Studies With TE-RAVs: Participants who previously participated in treatment studies in which boceprevir was administered were subsequently enrolled in Part 1 of the current follow-up study P05063 (NCT00689390). Participants may have received boceprevir or control peginterferon plus ribavirin (PR) in the previous treatment study. No treatment was administered in the current follow-up study.
- Participants From Narlaprevir Studies With TE-RAVs: Participants who previously participated in treatment studies in which narlaprevir was administered were subsequently enrolled in Part 2 of the current follow-up study P05063 (NCT00689390). Participants may have received narlaprevir or control PR in the previous treatment study. No treatment was administered in the current follow-up study.
Arm/Group | Participants From Boceprevir Studies With TE-RAVs | Participants From Narlaprevir Studies With TE-RAVs
Number analyzed (Participants) | 308 | 0
participants
  V36A TE-RAVs detected | 6 |
  __V36A TE-RAVs returned to WT (out of 6) | 6 |
  V36G TE-RAVs detected | 1 |
  __V36G TE-RAVs returned to WT (out of 1) | 1 |
  V36L TE-RAVs detected | 9 |
  __V36L TE-RAVs returned to WT (out of 9) | 8 |
  V36M TE-RAVs detected | 142 |
  __V36M TE-RAVs returned to WT (out of 142) | 135 |
  F43C TE-RAVs detected | 3 |
  __F43C TE-RAVs returned to WT (out of 3) | 3 |
  T54A TE-RAVs detected | 40 |
  __T54A TE-RAVs returned to WT (out of 40) | 40 |
  T54C TE-RAVs detected | 2 |
  __T54C TE-RAVs returned to WT (out of 2) | 2 |
  T54S TE-RAVs detected | 143 |
  __T54S TE-RAVs returned to WT (out of 143) | 104 |
  V55A TE-RAVs detected | 5 |
  __V55A TE-RAVs returned to WT (out of 5) | 3 |
  V107I TE-RAVs detected | 3 |
  __V107I TE-RAVs returned to WT (out of 3) | 2 |
  R155K TE-RAVs detected | 183 |
  __R155K TE-RAVs returned to WT (out of 183) | 154 |
  R155T TE-RAVs detected | 22 |
  __R155T TE-RAVs returned to WT (out of 22) | 20 |
  A156S TE-RAVs detected | 37 |
  __A156S TE-RAVs returned to WT (out of 37) | 35 |
  A156T TE-RAVs detected | 4 |
  __A156T TE-RAVs returned to WT (out of 4) | 4 |
  V158I TE-RAVs detected | 18 |
  __V158I TE-RAVs returned to WT (out of 16) | 16 |
  V158M TE-RAVs detected | 1 |
  __V158M TE-RAVs returned to WT (out of 1) | 1 |
  D168N TE-RAVs detected | 12 |
  __D168N TE-RAVs returned to WT (out of 12) | 11 |
  I170T TE-RAVs detected | 3 |
  __I170T TE-RAVs returned to WT (out of 3) | 3 |
  V170A TE-RAVs detected | 27 |
  __V170A TE-RAVs returned to WT (out of 27) | 24 |
  M175L TE-RAVs detected | 5 |
  __M175L TE-RAVs returned to WT (out of 5) | 2 |

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Reported During the LTFU
Description: Long-term safety was assessed based on the SAEs reported during the LTFU period. An SAE was any adverse drug or biologic or device experience occurring at any dose that resulted in any of the following outcomes: death, life-threatening AE, persistent or significant disability/incapacity, required in-patient hospitalization or prolongs hospitalization, congenital anomaly or birth defect. Important medical events that did not result in any of these outcomes could still be considered SAEs if they jeopardized the participant and/or required medical/surgical intervention, based on appropriate medical judgment. Grade 4 laboratory abnormalities and out of normal range liver function tests that were not accompanied by clinical manifestations were NOT considered SAEs.
Time Frame: From enrollment in the LTFU study to the last available date in the LTFU study (up to 3 years)
Population: All enrolled participants were included in safety analyses.
Measure: Number; unit: participants
Arm/Group | Participants From Boceprevir Studies | Participants From Narlaprevir Studies
Number analyzed (Participants) | 1907 | 47
participants | 136 | 2

5. Primary Outcome: Number of Participants That Discontinued the LTFU Due to SAEs
Description: An SAE was any adverse drug or biologic or device experience occurring at any dose that resulted in any of the following outcomes: death, life-threatening AE, persistent or significant disability/incapacity, required in-patient hospitalization or prolongs hospitalization, congenital anomaly or birth defect. Important medical events that did not result in any of these outcomes could still be considered SAEs if they jeopardized the participant and/or required medical/surgical intervention, based on appropriate medical judgment. Grade 4 laboratory abnormalities and out of normal range liver function tests that were not accompanied by clinical manifestations were NOT considered SAEs.
Time Frame: From enrollment in the LTFU study to the last available date in the LTFU study (up to 3 years)
Population: All enrolled participants were included in safety analyses.
Measure: Number; unit: participants
Arm/Group | Participants From Boceprevir Studies | Participants From Narlaprevir Studies
Number analyzed (Participants) | 1907 | 47
participants | 19 | 0

ADVERSE EVENTS:
Time Frame: From enrollment in the LTFU study to the last available date in the LTFU study (up to 3 years)
Description: As specified in the protocol, only serious adverse events (SAEs) were collected. Other Adverse Events were not monitored and not collected, thus no participants were at risk for these events. All enrolled participants were included in safety analyses.
Arm/Group | Participants From Boceprevir Studies | Participants From Narlaprevir Studies
Serious Adverse Events (participants affected / at risk) | 136/1907 | 2/47
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants From Boceprevir Studies (N=1907) | Participants From Narlaprevir Studies (N=47)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (2) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 (5) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 9 (9) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (2) | 0 (0)
ENDOCARDIAL FIBROELASTOSIS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HUNTINGTON'S DISEASE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0)
CORNEAL OEDEMA (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HERNIAL EVENTRATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PALATAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 2 (3) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 (2) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 4 (4) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 5 (5) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
ACUTE HEPATITIS B (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS PERFORATED (Infections and infestations) | 2 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (3) | 0 (0)
HEPATITIS C (Infections and infestations) | 1 (1) | 0 (0)
HERPES SIMPLEX PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RETINITIS (Infections and infestations) | 1 (2) | 0 (0)
SEPSIS (Infections and infestations) | 3 (3) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 2 (2) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
STAB WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ANAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIOLOALVEOLAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (11) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF HEAD AND NECK (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ARACHNOID CYST (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
TENSION HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0)
UTEROVAGINAL PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 2 (2) | 0 (0)
FINGER AMPUTATION (Surgical and medical procedures) | 1 (1) | 0 (0)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (2) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
LIVER TRANSPLANT (Surgical and medical procedures) | 1 (1) | 0 (0)
SHOULDER ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
VALVULOPLASTY CARDIAC (Surgical and medical procedures) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) agrees to provide to the sponsor 30 days prior to submission for publication or presentation, review results communications. Sponsor shall have editorial rights with respect to results communications and the right to review and comment on the data analysis and presentation with regard to proprietary information, the accuracy of the information contained in the publication, and to ensure that the presentation is fairly balanced and in compliance with FDA regulations.